CLINICAL TRIAL: NCT07250958
Title: Dome-Only Aneurysm Coiling in Severe Aneurysmal Subarachnoid Hemorrhage Observational Study
Brief Title: Dome-Only Aneurysm Coiling in Severe Aneurysmal Subarachnoid Hemorrhage
Acronym: DOME
Status: Not yet recruiting | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Akshitkumar MIstry, Assistant Professor Term, University of Louisville
Other Study IDs: 25.0321
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The DOME study is a clinical trial exploring a new treatment approach for patients who suffered a severe brain bleed due to an aneurysm.

DETAILED DESCRIPTION:
To prospectively capture data of patients treated with the guideline-recommended, standard-of-care dome-protection approach. The data will be used to determine:

* (Primary) Incidence of aneurysm re-rupture by 90 days, censored at the time of definitive aneurysm treatment or death, detected on a surveillance head CT or one obtained after a neurological decline.
* (Secondary) Measure functional status of patients around 90 days (+/- 14 days)
* (Secondary) Measure success of dome protection as determined by angiographic criteria and procedural complications

DOME protection is a treatment approach for patients who suffered a severe brain bleed due to an aneurysm. Instead of performing immediate, extensive surgery, this study investigates a minimally invasive procedure called "dome protection", which involves placing tiny coils to patch the most fragile part of the aneurysm. This method aims to prevent re-bleeding and allow the patient to stabilize before undergoing full aneurysm repair. The findings could lead to improved health outcomes in patients with aneurysmal subarachnoid hemorrhage by reducing procedure-related risks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* CT confirmed aSAH with an angiographically detected aneurysm
* World Federation of Neurological Sciences (WFNS) aSAH grade 3-5 aneurysm
* LAR available and gives consent within 72 hours after the onset of aSAH (or last known normal

Exclusion Criteria:

* Patients whose aneurysm judged appropriate for balloon-assisted coiling
* Patients whose aneurysm is bleeding from the "neck"
* Patients who are clinically judged to suffer imminent death within 24 hours.
* Pregnancy or positive urine pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with CT confirmed aSAH with an angiographically detected aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Re-rupture incidence | From procedure to 90-days post procedure.
  Detected on head CT

SECONDARY OUTCOMES:
Functional Outcome | 90 days (+-14 days) post procedure
  Measured on Modified Rankin Scale (MRS) Scored 0-6 where 0-No disability, 1=no significant disability, 2= slight disability, 3=moderate disability, 4=moderately severe disability, 5=severe disability, 6=dead. The higher the score the worse the outcome.
Accomplishment of Dome protection | From procedure through 90-days post procedure
  Based on angiographic goals: 1) partial coil obliteration of the aneurysm dome or increased contrast stasis within the aneurysm dome compared to pre-embolization angiography, 2) filling of the aneurysm neck, 3) no filling of the aneurysm dome wall, and 4) no filling of the aneurysm rupture site or extra-aneurysmal contrast extravasation.
Procedural complications during the dome-protection and delayed final procedures on the aneurysm | Time of procedure through 90 days post procedure
  Collection of adverse events.